CLINICAL TRIAL: NCT00732589
Title: Suprascapular Nerve Block in Hemiplegic Shoulder Pain.
Brief Title: SSNB in Hemiplegic Shoulder Pain
Acronym: SSNB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Jariya Boonhong/ Department of Rehabilitation Medicine, Faculty of Medicine, Chulalongkorn University, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chulalongkorn University
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2008-08

CONDITIONS: Shoulder Pain; Stroke
Keywords: suprascapular nerve block; shoulder pain; hemiplegia
MeSH Terms: conditions — Shoulder Pain; Stroke; Hemiplegia | interventions — Lidocaine; High-Energy Shock Waves; Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Suprascapular nerve block
  Interventions: Drug: 1% xylocaine
- B (Experimental): therapeutic ultrasound
  Interventions: Other: ultrasound

INTERVENTIONS:
Drug: 1% xylocaine — 10 cc. of 1%xylocaine, once a week
  Other Names: suprascapular nerve block
  Arms: A
Other: ultrasound — ultrasound at shoulder area about 10 mins.
  Other Names: therapeutic ultrasound
  Arms: B

SUMMARY:
The purpose of this study is to compare suprascapular nerve block with therapeutic ultrasound in stroke patients who have shoulder pain in weak side.

DETAILED DESCRIPTION:
Shoulder pain is a common complication after a cerebrovascular accident.Hemiplegic shoulder pain has been shown to affect stroke outcome in a negative way.It interferes with recovery after stroke:it can cause distress and reduced activities and can markedly hinder rehabilitation.Suprascapular nerve block has been shown to be effective as an analgesic for different indications such as shoulder capsulitis.The purpose of this study was to evaluate the effectiveness of this technique conjunction with a rehabilitation program to reduce shoulder pain in hemiplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients who develope shoulder pain at weak limb.
* Good conscious and able to access pain score.
* No history of drug reaction with xylocaine
* No history of fracture,tumor or blood tendency.
* Willing to enrolled to study and signs inform consent.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
VAS score of pain | 4 weeks after intervention

SECONDARY OUTCOMES:
Range of motion of the shoulder joint | 4 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jariya Boonhong, physiatist, Principal Investigator — Unaffiliation
Locations (1):
- Department of physical medicine and rehabilitation, Faculty of medicien, Chulalongkorn University, Bangkok, Bangkok, Thailand